CLINICAL TRIAL: NCT03456531
Title: Effect of Pulsed Radiofrequency to the Suprascapular Nerve in Treating Frozen Shoulder Pain
Brief Title: Pulsed Radiofrequency for Frozen Shoulder Chronic Pain (PRFFSCP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmeen alaa-eldeen elmasry, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSN PRF
Record Dates: First submitted 2018-02-24; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Pulsed Radiofrequency Treatment; Aspirin; Analgesics

STUDY DESIGN:
Intervention Model Description: prospective randomized clinically controlled study .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): 20 patients will receive pulsed radiofrequency for 6 minutes to suprascapular nerve
  Interventions: Device: pulsed radiofrequency
- group 2 (Placebo Comparator): 20 patients will receive their medical treatment in the form of NSAIDs "ibubrofen,Aspirin"
  Interventions: Drug: NSAIDs "ibubrofen,Aspirin"

INTERVENTIONS:
Device: pulsed radiofrequency — The patient will have pulsed radiofrequency to suprascapular nerve for 6 minutes
  Other Names: PRF
  Arms: group 1
Drug: NSAIDs "ibubrofen,Aspirin" — medical treatment as NSAIDs "ibubrofen,Aspirin"
  Other Names: Analgesics
  Arms: group 2

SUMMARY:
this study to detect the effect of pulsed radiofrequency to the suprascapular nerve in treating chronic pain and to evaluate range of motion of shoulder joint after the intervention

DETAILED DESCRIPTION:
Adhesive capsulitis (also known as frozen shoulder) is a painful and disabling disorder of unclear cause in which the shoulder capsule, the connective tissue surrounding the glenohumeral joint of the shoulder, becomes inflamed and stiff, greatly restricting motion and causing chronic pain. Pain is usually constant, worse at night, and with cold weather. Certain movements or bumps can provoke episodes of tremendous pain and cramping. The condition is thought to be caused by injury or trauma to the area and may have an autoimmune component.

Frozen shoulder patients usually present in the sixth decade of life, and onset before the age of 40 is very uncommon. The peak age is 56, and the condition occurs slightly more often in women than men In 6-17% of patients, the other shoulder becomes affected, usually within five years, and after the first has resolved .The non-dominant shoulder is slightly more likely to be affected. Few attempts have been made to calculate the cumulative lifetime risk of frozen shoulder. In the Scandinavian population at risk, it has been estimated at a minimum of 2% per year. Recurrence is highly unusual.Frozen shoulder can be a primary or idiopathic problem or it may be associated with another systemic illness. By far the most common association of a secondary frozen shoulder is diabetes mellitus. The incidence of frozen shoulder in diabetes patients is reported to be 10%-36%. The incidence in type 1 and type 2 diabetes is similar.Unfortunately, frozen shoulder in diabetes is often more severe and is more resistant to treatment . The natural history of the diabetic painful stiff shoulder and found a restriction in the range of motion in 35 (65%) of 54 shoulders at a mean follow-up of 29 months . There is an association with Dupuytren's disease in the hand, proposing that the contracting shoulder tissue itself represents a form of fibromatosis . Much more rarely, secondary frozen shoulder may be associated with conditions such as hyperthyroidism hypothyroidism and hypoadrenalism. Additional associations include Parkinson's disease, cardiac disease, pulmonary disease, and stroke although the pathological condition here may be different from idiopathic frozen shoulder. Clearly, in the case of stroke, shoulder stiffness may be simply the result of muscle spasticity in the shoulder region.Frozen shoulder has also been reported subsequent to non-shoulder surgical procedures, such as cardiac surgery cardiac catheterisation through the brachial artery neurosurgery and radical neck dissection .

The stages of frozen shoulder are 3 stages Freezing In the "freezing" stage, the patient slowly has more and more pain. As the pain worsens, the shoulder loses range of motion. Freezing typically lasts from 6 weeks to 9 months.

Frozen Painful symptoms may actually improve during this stage, but the stiffness remains. During the 4 to 6 months of the "frozen" stage, daily activities may be very difficult.

Thawing Shoulder motion slowly improves during the "thawing" stage. Complete return to normal or close to normal strength and motion typically takes from 6 months to 2 years.

Movement of the shoulder is severely restricted, with progressive loss of both active and passive range of motion The condition is sometimes caused by injury, leading to lack of use due to pain, but also often arises spontaneously with no obvious preceding trigger factor (idiopathic frozen shoulder). Rheumatic disease progression and recent shoulder surgery can also cause a pattern of pain and limitation similar to frozen shoulder. Intermittent periods of use may cause inflammation.

One sign of a frozen shoulder is that the joint becomes so tight and stiff that it is nearly impossible to carry out simple movements, such as raising the arm. The movement that is most severely inhibited is external rotation of the shoulder.

In frozen shoulder, there is a lack of synovial fluid, which normally helps the shoulder joint, a ball and socket joint, move by lubricating the gap between the humerus(upper arm bone) and the socket in the shoulder blade. The shoulder capsule thickens, swells, and tightens due to bands of scar tissue (adhesions) that have formed inside the capsule. As a result, there is less room in the joint for the humerus, making movement of the shoulder stiff and painful. This restricted space between the capsule and ball of the humerus distinguishes adhesive capsulitis from a less complicated, painful, stiff shoulder .

Frozen shoulder generally gets better over time, although it may take up to 3 years.The focus of treatment is to control pain and restore motion and strength through physical therapy.

Nonsurgical Treatment More than 90% of patients improve with relatively simple treatments to control pain and restore motion.

Non-steroidal anti-inflammatory medicines. Drugs like aspirin and ibuprofen reduce pain and swelling.

Steroid injections. Cortisone is a powerful anti-inflammatory medicine that is injected directly into shoulder joint.

Physical therapy. Specific exercises will help restore motion. These may be under the supervision of a physical therapist or via a home program. Therapy includes stretching or range of motion exercises for the shoulder. Sometimes heat is used to help loosen the shoulder up before the stretching exercises.

Surgical Treatment If symptoms are not relieved by therapy and anti-inflammatory medicines, surgery may be considered.

The goal of surgery for frozen shoulder is to stretch and release the stiffened joint capsule. The most common methods include manipulation under anesthesia and shoulder arthroscopy.

Manipulation under anesthesia. During this procedure shoulder will be forced to move which causes the capsule and scar tissue to stretch or tear. This releases the tightening and increases range of motion Shoulder arthroscopy. In this procedure, the surgeon will cut through tight portions of the joint capsule. This is done using pencil-sized instruments inserted through small incisions around the shoulder In many cases, manipulation and arthroscopy are used in combination to obtain maximum results. Most patients have very good outcomes with these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are complaining of chronic pain due to frozen shoulder for more than 3 weeks.
* All of them will be above 30 years and from areas nearby our hospital to make the follow up easy and complete.
* All participants will be ASA physical status I-III and random blood glucose will be measured 1 week before intervention.

Exclusion Criteria:

* Those with infection at site of injection, coagulopathy or other bleeding diathesis, pre-existing neurologic deficit in targeted region, those with history of chronic opioid use and those who refused to participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
pain measure | 1 week
  to evaluate the efficacy of pulsed radiofrequency lesioning to the suprascapular nerve in treating pain in frozen shoulder using numeric pain rating scale where 0 is no pain and 10 is the worst pain ever

SECONDARY OUTCOMES:
Range of motion of the shoulder | 3 months
  evaluate patient range of motion after the intervention using the simple shoulder test "by answering 12 questions "

CONTACTS AND LOCATIONS:
Overall Officials: ayman othman, proffessor, Study Director — Assiut univerisity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liliang PC, Lu K, Liang CL, Tsai YD, Hsieh CH, Chen HJ. Pulsed radiofrequency lesioning of the suprascapular nerve for chronic shoulder pain: a preliminary report. Pain Med. 2009 Jan;10(1):70-5. doi: 10.1111/j.1526-4637.2008.00543.x. PMID 19222771
- [Background] Jang JS, Choi HJ, Kang SH, Yang JS, Lee JJ, Hwang SM. Effect of pulsed radiofrequency neuromodulation on clinical improvements in the patients of chronic intractable shoulder pain. J Korean Neurosurg Soc. 2013 Dec;54(6):507-10. doi: 10.3340/jkns.2013.54.6.507. Epub 2013 Dec 31. PMID 24527194